CLINICAL TRIAL: NCT04563325
Title: Oral-only Antibiotics for Bone and Joint Infections in Children - A Nationwide Randomized Controlled Trial
Brief Title: Oral-only Antibiotics for Bone and Joint Infections in Children
Acronym: CHILD@HOME_BJI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The research foundation of Copenhagen University Hospital, Rigshospitalet (Unknown); Copenhagen Health Science Partners (Unknown); Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Allan Bybeck Nielsen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20009117
Record Dates: First submitted 2020-09-13; First posted 2020-09-24 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Osteomyelitis; Septic Arthritis; Bone Infection; Joint Infection; Bone and Joint Infection
MeSH Terms: conditions — Osteomyelitis; Arthritis, Infectious | interventions — Amoxicillin-Potassium Clavulanate Combination; Dicloxacillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor (qualified pediatrician or pediatric surgeon) of the primary endpoint (sequelae 6 months after initiation of treatment) will be blinded for the intervention as well as any other details on the course of disease. The assessor will be informed about the age of the child as well as the approximate location of the infection and will perform a predefined systematic clinical examination of the relevant area (categories: 1) lower extremities, 2) upper extremities incl. claviculae and scapulae and 3) columna, costae and sternum). The exact anatomical location including side (left or right) will not be revealed. The child and parents will be followed by a study nurse who will secure that the blinding is respected. The primary endpoint is met if there are any positive findings related to the previously infected bone or joint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): < 5 years: High-dose oral co-amoxiclav (1:8) 33 mg amoxicillin/kg/dose (max. 1 g) three-times daily (TDS) until clinical and paraclinical improvement (min. 3 days) followed by oral co-amoxiclav (1:4) 17 mg amoxicillin/kg/dose (max. 500 mg) TDS for 7 days (arthritis) or 21 days (osteomyelitis).
  =/> 5 years: High-dose oral dicloxacillin 50 mg/kg/dose (max. 2 g) four-times daily (QID) until clinical and paraclinical improvement (min. 3 days) followed by oral dicloxacillin 25 mg/kg/dose (max. 1 g) QID for 7 days (arthritis) or 21 days (osteomyelitis).
  Treatment will be adjusted according to microbiological findings.
  Interventions: Drug: Oral co-amoxiclav or oral dicloxacillin only
- Standard (Active Comparator): IV ceftriaxon 100 mg/kg/dose (max. 4 g) once daily (QD) (all ages) until clinical and paraclinical improvement (min. 3 days) followed by:
  < 5 years: Oral co-amoxiclav (1:4) 17 mg amoxicillin/kg/dose (max. 500 mg) TDS for 7 days (arthritis) or 21 days (osteomyelitis).
  >/= 5 years: Oral dicloxacillin 25 mg/kg/dose (max. 1 g) QID for 7 days (arthritis) or 21 days (osteomyelitis).
  Treatment will be adjusted according to microbiological findings.
  Interventions: Drug: IV ceftriaxon followed by oral co-amoxiclav or oral dicloxacillin

INTERVENTIONS:
Drug: Oral co-amoxiclav or oral dicloxacillin only — High dose oral treatment followed by standard dose oral treatment
  Arms: Experimental
Drug: IV ceftriaxon followed by oral co-amoxiclav or oral dicloxacillin — IV treatment followed by standard dose oral treatment
  Arms: Standard

SUMMARY:
A nationwide, multicenter, randomized, non-inferiority trial of children with bone and joint infections. The primary objective is to determine if oral-only antibiotics (experimental arm) is non-inferior to initial intravenous antibiotics followed by oral therapy (control arm). Children will be randomized 1:1. The total treatment duration is identical in both groups. The study is open label with blinding of the primary endpoint assessor.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 months to 18 years with antibiotic treatment of uncomplicated bone or joint infection.

Exclusion Criteria:

1. Severe disease, e.g. septic shock, or any concomitant infection, e.g. necrotizing fasciitis, requiring IV antibiotics in the opinion of the treating clinician.
2. Complicated bone or joint infection, e.g. prosthetic material, infection secondary to or complicated by trauma, severe pyomyositis or other substantial soft tissue infections.
3. Expected need of major surgery within the first 24 hours of treatment, e.g. drilling, debridement, fenestration, surgical drainage, synovectomy. Minor surgery as diagnostic surgical bone biopsy or diagnostic joint fluid aspiration including lavage is not a criterion for exclusion.
4. Significant co-morbidities that might influence the choice of treatment or the course of the infection, e.g. immunodeficiency, immunosuppressive therapy, sickle cell anemia.
5. Previous bone or joint infection.
6. Antibiotic therapy for more than 24 hours before inclusion.
7. Documented pathogen with limited treatment options that do not permit randomization, e.g. the pathogen is only sensitive to intravenous antibiotics.
8. Prior enrolment in the trial

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Sequelae at 6 months | 6 months
  Proportion of children with sequelae 6 months after initiation of treatment defined as abnormal mobility or function of the affected joint/bone. Evaluated by blinded clinical examination by a qualified pediatrician and/or pediatric orthopedic surgeon.

SECONDARY OUTCOMES:
Non-acute treatment failure. | 28 days
  Proportion of children with change of antibiotic therapy due to non-acute treatment failure. This will be evaluated by two pediatric specialists and is suggested by e.g. 1) temperature above 38,5 after more than 72 hours of antibiotic therapy, 2) increasing CRP ( C-reactive protein) after more than 96 hours of antibiotic therapy and 3) no improvement in mobility or pain after 120 hours of antibiotic therapy.
Recurrent infection | 6 months
  Proportion of children with recurrence of symptoms and signs (same anatomical location) after completion of antibiotic treatment requiring further antibiotic administration

OTHER OUTCOMES:
Safety Outcome 1: Severe complications during antibiotic treatment. | 28 days
  Proportion of children with severe complications during antibiotic treatment, e.g. need for intensive care, septic shock, organ failure, pyomyositis, endocarditis, deep venous thrombosis.
Safety Outcome 2: Surgical intervention | 28 days
  Proportion of children with need for surgical intervention during antibiotic treatment. Diagnostic surgical intervention (diagnostic joint aspiration or diagnostic bone biopsy) excluded.
Safety Outcome 3: Treatment related adverse events | 3 months
  Proportion of children with treatment related adverse events e.g. complications of IV access (infection, need for replacement, extravasation) and drug side effects reported by medical staff or by parents (electronic questionnaire).
Time to apyrexia from initiation of antibiotic treatment | 28 days
Mobility and pain | 14 days
  Level of mobility and pain assessed by daily grading of symptoms by medical staff as well as daily standardized pain scores by participants and/or parents. Score systems: Visual Analog Scale (VAS) or Face Legs Activity Cry Consolability (FLACC) scale, both with scores from 0 (no pain) to 10 (worst pain). [14 days]
Total duration of antibiotic therapy | 3 months
Sequelae at 12 months | 12 months
  Proportion of children with sequelae, e.g. abnormal mobility, growth abnormalities assessed by clinical examination by a qualified pediatrician 12 month after initiation of treatment.
Radiological abnormalities at 12 months | 12 months
  Proportion of children with radiological abnormalities assessed by a qualified radiologist 12 months after the initiation of treatment.
Secondary infection | 3 months
  Proportion of children with secondary infection with antimicrobial-resistant organisms or Clostridium difficile

CONTACTS AND LOCATIONS:
Overall Officials: Allan Bybeck Nielsen, MD, Principal Investigator — Rigshospitalet, Denmark; Ulrikka Nygaard, Ass Prof PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be shared. The exact plan for sharing Individual Participant Data (IPD) is being prepared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Nielsen AB, Holm M, Lindhard MS, Glenthoj JP, Borch L, Hartling U, Schmidt LS, Rytter MJH, Rasmussen AH, Damkjaer M, Lemvik G, Petersen JJH, Sondergaard MJ, Thaarup J, Kristensen K, Jensen LH, Hansen LH, Lawaetz MC, Gottliebsen M, Horsager TH, Zaharov T, Hoffmann TU, Nygaard T, Justesen US, Stensballe LG, Vissing NH, Blanche P, Schmiegelow K, Nygaard U. Oral versus intravenous empirical antibiotics in children and adolescents with uncomplicated bone and joint infections: a nationwide, randomised, controlled, non-inferiority trial in Denmark. Lancet Child Adolesc Health. 2024 Sep;8(9):625-635. doi: 10.1016/S2352-4642(24)00133-0. Epub 2024 Jul 15. PMID 39025092
- [Derived] Bybeck Nielsen A, Borch L, Damkjaer M, Glenthoj JP, Hartling U, Hoffmann TU, Holm M, Helleskov Rasmussen A, Schmidt LS, Schmiegelow K, Stensballe LG, Nygaard U; Local Investigators. Oral-only antibiotics for bone and joint infections in children: study protocol for a nationwide randomised open-label non-inferiority trial. BMJ Open. 2023 Jun 1;13(6):e072622. doi: 10.1136/bmjopen-2023-072622. PMID 37263683

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04563325/SAP_001.pdf